CLINICAL TRIAL: NCT05626179
Title: A Mass Balance Study of [14C]IBI351 in Healthy Male Chinese Subjects
Brief Title: A Study of [14C]IBI351 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIBI351P002
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] IBI351 (Other): Recommended dose of [14C] IBI351
  Interventions: Drug: [14C] IBI351

INTERVENTIONS:
Drug: [14C] IBI351 — The oral formulation of [14C] IBI351 was formulated as a suspension for subjects to take orally in drinking water under fasting conditions

SUMMARY:
This study is to evaluate the mass balance of single oral dose of [14C] IBI351 in healthy subjects. Six to eight healthy male subjects were planned to be enrolled. After passing the screening, subjects were admitted to hospital and received training on medication, urine and feces collection and other procedures to ensure that they could perform relevant operations according to the protocol and SOP requirements. On the evening before medication, the patient had standard meals, and fasted uniformly overnight. On D1, the suspension containing recommended dose of [14C] IBI351 was administered in the morning on an empty stomach. Subjects have standardized meal during the trial and blood, urine, and feces samples were collected and safety laboratory tests were performed as scheduled.

ELIGIBILITY:
Inclusion Criteria：

1. Voluntarily sign the informed consent form before the trial, and fully understand the content, process and possible adverse reactions of the trial.
2. Healthy male subjects aged 18 to 45 years (including both ends) at the time of signing informed consent.
3. Body weight is not less than 50 kg, and body mass index (BMI) is in the range of 19 ~ 26 kg/m2 (including both ends).
4. Vital signs, physical examination, laboratory tests (including blood routine, urine routine, blood biochemistry, coagulation, etc.), chest radiography, 12-lead ECG and other results were unremarkable; or abnormal examination results but judged by the investigator as clinically insignificant.

Exclusion Criteria

1. allergic constitution; known hypersensitivity to any component of the test drug or its preparation.
2. have special requirements for diet and cannot abide by the unified diet; or lactose intolerance.
3. history of dysphagia or any gastrointestinal disease that affects drug absorption.
4. blood donation or massive blood loss (> 200 mL) within 3 months before screening, or blood transfusion within 1 month.
5. Have taken an investigational product or participated in any clinical trial within 3 months before taking the study drug.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
cumulative recovery of total radioactivity in excreta (urine and feces) | approximately 30 days after first dose
percentage of metabolite in total exposure AUC in plasma (% AUC) | approximately 30 days after first dose
percentage of each metabolite in urine to administered dose (% of administered dose) | approximately 30 days after first dose
Percentage of each metabolite in feces to administered dose (% of administered dose) | approximately 30 days after first dose
total radioactivity ratio for whole blood/plasma | approximately 30 days after first dose
maximum concentrations (Cmax ) for total plasma radioactivity | approximately 30 days after first dose
time-to-maximum concentration (Tmax) for total plasma radioactivity | approximately 30 days after first dose
half-life (t1/2) for total plasma radioactivity | approximately 30 days after first dose
area under the curve from time 0 to the last time point (AUC0-t) for total plasma radioactivityarea under the curve from time 0 to the last time point (AUC0-t) for total plasma radioactivity | approximately 30 days after first dose
area under the curve from time 0 to infinity(AUC0-inf) for total plasma radioactivity | approximately 30 days after first dose
apparent clearance (CL/F) for total plasma radioactivity | approximately 30 days after first dose
apparent volume of distribution(Vz/F) for total plasma radioactivity | approximately 30 days after first dose

SECONDARY OUTCOMES:
maximum concentrations (Cmax ) for plasma | approximately 30 days after first dose
time-to-maximum concentration (Tmax) for plasma | approximately 30 days after first dose
area under the curve from time 0 to the last time point (AUC0-t) for plasma | approximately 30 days after first dose
area under the curve from time 0 to infinity(AUC0-inf) for plasma | approximately 30 days after first dose
apparent clearance (CL/F) for plasma | approximately 30 days after first dose
apparent volume of distribution(Vz/F) for plasma | approximately 30 days after first dose
adverse events | approximately 30 days after first dose
abnormality in vital signs | approximately 30 days after first dose
abnormality in ECG parameters | approximately 30 days after first dose
abnormality in physical examination | approximately 30 days after first dose
abnormality in hematology parameters | approximately 30 days after first dose
abnormality in clinical chemistry parameters | approximately 30 days after first dose
abnormality in routine urinalysis parameters | approximately 30 days after first dose
abnormality in routine stool parameters | approximately 30 days after first dose
abnormality in coagulation parameters | approximately 30 days after first dose
abnormality in Troponin T (TnT) | approximately 30 days after first dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China